CLINICAL TRIAL: NCT06770491
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Phase 1 Study to Assess the Safety, Tolerability, and Pharmacokinetic Profiles of Y-3 in Healthy Adult Volunteers in the United States
Brief Title: A Phase 1 Study of Y-3 in US Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: Y-3-LC-06
Record Dates: First submitted 2024-12-24; First posted 2025-01-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Safety; Tolerability; Pharmacokinetic Study in Healthy Volunteers
Keywords: safety; tolerability; Pharmacokinetic study in healthy volunteers; Y-3; stroke
MeSH Terms: conditions — Stroke | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: CRA, sponsor，CRO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Y-3 for injection (Y-3) (Experimental): The investigational drug (Y-3) consists of two parts: Y-3 for injection (lyophilized powder) （20 mg）and Solvent for Y-3 for injection (concentrated solution)（3ml (containing 0.6 g propylene glycol)）.
  Subjects will receive Y-3 or placebo on the morning of the dosing day. Drinking water is prohibited from 1 hour before administration until the end of dosing, and subjects may have meals 4 hours after administration.
  Using a sterile syringe, withdraw dedicated solution into the lyophilized powder vial of Y-3 or placebo. Shake the vial manually until the powder is dissolved. Once completely dissolved, use a sterile syringe to transfer the solution into the infusion bottle (normal saline) and gently mix by swirling. The intravenous infusion volume is 250 ml, and infusion time is 60 min ± 10 min. The storage time of the reconstituted drug product or placebo should not exceed 4 hours at room temperature or 24 hours at refrigerated temperature prior to initiation of administration.
  Interventions: Drug: Y-3 for injection
- placebo (Placebo Comparator): The placebo consists of two parts: placebo (lyophilized powder) and Solvent for Y-3 for injection(concentrated solution).
  Subjects will receive Y-3 or placebo on the morning of the dosing day. Drinking water is prohibited from 1 hour before administration until the end of dosing, and subjects may have meals 4 hours after administration.
  Using a sterile syringe, withdraw dedicated solution into the lyophilized powder vial of Y-3 or placebo. Shake the vial manually until the powder is dissolved. Once completely dissolved, use a sterile syringe to transfer the solution into the infusion bottle (normal saline) and gently mix by swirling. The intravenous infusion volume is 250 ml, and infusion time is 60 min ± 10 min. The storage time of the reconstituted drug product or placebo should not exceed 4 hours at room temperature or 24 hours at refrigerated temperature prior to initiation of administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Y-3 for injection — The investigational drug (Y-3) consists of two parts: Y-3 for injection (lyophilized powder) and Solvent for Y-3 for injection (concentrated solution).
  Name: Y-3 for injection Strength: 20 mg Dosage Form: Lyophilized powder for injection Storage Condition: 2-8°C Supplier: Neurodawn Pharmaceutical Co., Ltd. Name: Reconstitution diluent for Y-3 for injection Strength: 3ml (containing 0.6 g propylene glycol) Dosage Form: Concentrated solution for injection Storage Condition: 2-8°C Supplier: Neurodawn Pharmaceutical Co., Ltd.
  Arms: Y-3 for injection (Y-3)
Drug: Placebo — The placebo consists of two parts: placebo (lyophilized powder) and Solvent for Y-3 for injection(concentrated solution).
  Name: Placebo Strength: 0 mg Dosage Form: Lyophilized powder for injection Storage Condition: 2-8°C Supplier: Neurodawn Pharmaceutical Co., Ltd. Name: Solvent for Y-3 for injection Strength: 3 mL (containing 0.6 g propylene glycol) Dosage Form: Concentrated solution for injection Storage Condition: 2-8°C Supplier: Neurodawn Pharmaceutical Co., Ltd.
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability, and pharmacokinetic profiles of Y-3 in healthy adult volunteers in the United States. The main questions it aims to answer are:

* What the pharmacokinetic profiles of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers?
* If drug Y-3 (40mg and 60 mg) is safe and tolerate in the US healthy adult volunteers.

Researchers will compare drug Y-3 (40 mg and 60 mg) to a placebo (a look-alike substance that contains no drug) to see what the pharmacokinetic profiles of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers and if drug Y-3 (40mg and 60 mg) is safe and tolerate in the US healthy adult volunteers.

Participants will:

* Take drug Y-3 (40 mg) or Y-3 (60 mg) or a placebo only once.
* Answer questions regarding your medical history.
* Comply with the study procedures and requests.
* Complete all tests and collections of PK Sampling.
* Must not have any special dietary requirements and be able to consume the food (low-fat) provided by Tranquil Clinical Research during your 4-night stay.
* Must avoid excessive ( > 8 cups per day) caffeine consumption (i.e. coffee or tea) during your time in the study.
* Must not consume any food or beverage rich in grapefruit, papaya, or mango during your time in the study.
* Must not take any other medications, including traditional Chinese medicines and herbal medicines, during your time in the study.
* Must avoid sexual activity or use non-drug contraceptive measures (i.e. condoms) during your time in the study.
* Female participants must not become pregnant while in the study.
* Must not receive any vaccinations during your time in the study.
* Must not donate blood for purposes outside of study procedures during your time in the study.
* Must not drink alcohol during your time in the study.
* Must not smoke during your time in the study.
* Inform your Study Doctor if you no longer wish to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Medically documented as healthy at the time of screening as determined by their medical history, medical assessment, physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory tests, etc.
2. Within 18-45 years at the time of informed consent, inclusive.
3. Body weight ≥ 50 kg for male and ≥ 45 kg for female, body mass index (BMI) within the range of 19 - 28 kg/m2, inclusive.
4. Fully understand and provide a signed informed consent before performing any study-related procedures.
5. Comply with the study and follow-up procedures.

Exclusion Criteria:

1. Known allergy to Y-3 or any of its excipients.
2. Have disease history or current disease that may affect the safety evaluation of the subject or the internal process of the study drug, that the investigator judged to be of clinical significance, including the cardiovascular system, endocrine system, central nervous system, digestive system, respiratory system, hematological system, immunology, psychiatry, metabolic abnormalities, etc.
3. Clinically significant abnormal 12-lead electrocardiograms (ECG) and vital signs judged by the investigator.
4. Clinically significant abnormal laboratory tests (hematology, serum chemistry, coagulation, urinalysis, etc.) and other screening tests judged by the investigator.
5. Test positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, syphilis antibody or human immunodeficiency virus (HIV) antibody.
6. Alcoholics or regular drinkers within 6 months prior to screening, that is, those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of alcohol with 40% alcohol content or 150 mL of wine), or whose alcohol breath test results are greater than 0.0 mg/100 mL, or who cannot abstain from alcohol during the study.
7. Smokers, that is, those who smoke more than 3 cigarettes per day within 3 months prior to screening, or those who cannot comply with the prohibition of smoking during the study.
8. Current or former drug users, or positive urine screen for drugs of abuse at screening.
9. Have special requirements for diet and cannot follow the unified diet.
10. Drink too much tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup = 250 mL) every day within 3 months prior to screening, or who have consumed any diet (food or beverage) rich in grapefruit, pitaya and mango within 14 days prior to screening.
11. Have taken any prescription drug or over-the-counter drug, traditional Chinese medicine or herbal medicine, health products within 14 days prior to screening, or 5 half-lives, whichever is longer, before the first dose of study drug, or have received vaccine inoculation within 14 days prior to screening; or plan to inoculate vaccine during the study.
12. Participated in any other clinical trials within 3 months prior to screening.
13. Donation or loss of blood equal to or in excess of 200 mL within 3 months prior to screening.
14. Female subjects who have unprotected intercourse within 14 days prior to screening, or pregnant or lactating women.
15. Male subjects (or their partners) or female subjects have baby plans during the whole trial period and within 3 months after the end of the trial, or subjects are unwilling to take one or more non-drug contraceptive measures (such as complete abstinence, condoms, ligation, etc.) during the study.
16. Subjects voluntarily withdraw from the study due to personal reason, or subjects who the investigator believes are not suitable for enrollment for other reasons.
17. Suicidal ideation, history of suicidal behavior, or history of psychiatric comorbidities.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the Cmax of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin | treatment period (Day1-Day4)
  Maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the AUC 0-t of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
  Calculated according to linearity trapezoidal rule:
  AUC (i, i+1) = (Ti+1-Ti) (Ci+Ci+1) /2, and AUC0-t is the sum of all AUC (i, i + 1).
Evaluate the AUC 0-∞ of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Area under the concentration-time curve from time 0 to infinity (extrapolated). AUC 0-∞ =AUC 0-t + Ct/λz (Ct is the last measured plasma concentration).
Evaluate the Tmax of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Time to reach maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the t1/2 of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Terminal elimination half-life. t1/2 = ln2/λ。
Evaluate the λz of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
Evaluate the AUC_%Extrap of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
Evaluate the Vz of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Volume of distribution. Vz = Div/AUC0-∞/λz
Evaluate the CL of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Total body clearance. CLz = Div /AUC0-∞
Evaluate the MRT 0-t of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Mean residence time within the time from time zero to the lowest testing plasma concentration. MRT0-t = AUMC0-t/AUC0-t.
Evaluate the MRT 0-∞ of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by venous blood and Phoenix WinNonlin. | treatment period (Day1-Day4)
  Mean residence time extrapolated from zero to infinity. MRT 0-∞ = AUMC 0-∞/AUC 0-∞.

SECONDARY OUTCOMES:
Evaluate the safety of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of physical examinations after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation.
Evaluate the safety of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of vital signs after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature） will be assessed by according equipments.(electronic sphygmomanometer，thermometer).
Evaluate the safety of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of 12-lead ECG after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the safety of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of laboratory tests after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the safety of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by the rates of adverse events after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe".
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Evaluate the tolerability of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of physical examinations after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through obeservation.
Evaluate the tolerability of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of vital signs after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature） will be assessed by according equipment.(electronic sphygmomanometer，thermometer).
Evaluate the tolerability of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of 12-lead ECG after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the tolerability of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by Incidence of subject getting abnormal results of laboratory tests after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the tolerability of single ascending doses of Y-3 (40 mg and 60 mg) in the US healthy adult volunteers by the rates of adverse events after treatment. | This study comprises a screening period (Day -14 to Day -2), a baseline period (Day -1), a treatment period (Day1 - Day4), and a safety follow-up period (Day7).
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment. The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of "mild", "moderate" and "severe". The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.

CONTACTS AND LOCATIONS:
Locations (1):
- Tranquil Clinical Research, Webster, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hill MD, Goyal M, Menon BK, Nogueira RG, McTaggart RA, Demchuk AM, Poppe AY, Buck BH, Field TS, Dowlatshahi D, van Adel BA, Swartz RH, Shah RA, Sauvageau E, Zerna C, Ospel JM, Joshi M, Almekhlafi MA, Ryckborst KJ, Lowerison MW, Heard K, Garman D, Haussen D, Cutting SM, Coutts SB, Roy D, Rempel JL, Rohr AC, Iancu D, Sahlas DJ, Yu AYX, Devlin TG, Hanel RA, Puetz V, Silver FL, Campbell BCV, Chapot R, Teitelbaum J, Mandzia JL, Kleinig TJ, Turkel-Parrella D, Heck D, Kelly ME, Bharatha A, Bang OY, Jadhav A, Gupta R, Frei DF, Tarpley JW, McDougall CG, Holmin S, Rha JH, Puri AS, Camden MC, Thomalla G, Choe H, Phillips SJ, Schindler JL, Thornton J, Nagel S, Heo JH, Sohn SI, Psychogios MN, Budzik RF, Starkman S, Martin CO, Burns PA, Murphy S, Lopez GA, English J, Tymianski M; ESCAPE-NA1 Investigators. Efficacy and safety of nerinetide for the treatment of acute ischaemic stroke (ESCAPE-NA1): a multicentre, double-blind, randomised controlled trial. Lancet. 2020 Mar 14;395(10227):878-887. doi: 10.1016/S0140-6736(20)30258-0. Epub 2020 Feb 20. PMID 32087818
- [Result] Chamorro A, Lo EH, Renu A, van Leyen K, Lyden PD. The future of neuroprotection in stroke. J Neurol Neurosurg Psychiatry. 2021 Feb;92(2):129-135. doi: 10.1136/jnnp-2020-324283. Epub 2020 Nov 4. PMID 33148815
- [Result] Campbell BCV, De Silva DA, Macleod MR, Coutts SB, Schwamm LH, Davis SM, Donnan GA. Ischaemic stroke. Nat Rev Dis Primers. 2019 Oct 10;5(1):70. doi: 10.1038/s41572-019-0118-8. PMID 31601801
- [Result] Wu H, Huang Z, Wang X, Chen M, Chen W, Hua Y, Ren J, Shen L, Song Y, Zhou Y, Luo C, Lin Y, Wang Y, Chang L, Li F, Zhu D. Preclinical evaluation of ZL006-05, a new antistroke drug with fast-onset antidepressant and anxiolytic effects. Stroke Vasc Neurol. 2023 Dec 29;8(6):463-474. doi: 10.1136/svn-2022-002156. PMID 37185136
- [Result] Xu X, Chen M, Zhu D. Reperfusion and cytoprotective agents are a mutually beneficial pair in ischaemic stroke therapy: an overview of pathophysiology, pharmacological targets and candidate drugs focusing on excitotoxicity and free radical. Stroke Vasc Neurol. 2024 Aug 27;9(4):351-359. doi: 10.1136/svn-2023-002671. PMID 37832977
- [Result] Fisher M; Stroke Therapy Academic Industry Roundtable. Recommendations for advancing development of acute stroke therapies: Stroke Therapy Academic Industry Roundtable 3. Stroke. 2003 Jun;34(6):1539-46. doi: 10.1161/01.STR.0000072983.64326.53. Epub 2003 May 15. PMID 12750546
- [Result] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721